CLINICAL TRIAL: NCT02085551
Title: The Prism Trial: A Retrospective Case Review of Technical Success Using the Penumbra and Indigo Systems for Mechanical Thrombectomy in the Periphery
Brief Title: Case Review of the Penumbra and Indigo Systems for Mechanical Thrombectomy in the Periphery
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 7051
Record Dates: First submitted 2014-03-05; First posted 2014-03-13 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Peripheral Arterial Occlusion or Emboli
Keywords: peripheral arterial occlusion; visceral emboli; limb ischemia; adverse events; Indigo System; aspiration; mechanical thrombectomy
MeSH Terms: conditions — Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mechanical thrombectomy by the Indigo System (Experimental)
  Interventions: Device: Mechanical Thrombectomy by the Indigo System

INTERVENTIONS:
Device: Mechanical Thrombectomy by the Indigo System

SUMMARY:
The primary objective of this retrospective case review study is to determine the safety and effectiveness of the Penumbra and Indigo Systems for mechanical thrombectomy in a cohort of patients with confirmed peripheral or visceral arterial occlusion or embolus. This is a retrospective, single arm, multi-center trial. Up to 100 patients at up to 10 centers will be enrolled. Angiographic assessment of vessel patency at immediate post-procedure as measured by TIMI scores and procedural serious adverse events are assessed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a peripheral or visceral arterial occlusion or embolus (TIMI 0-1) prior to treatment.
* Treatment with components of the Penumbra and/or Indigo System.

Exclusion Criteria:

* Participation in another clinical investigation that may confound the results of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saxon, MD, Principal Investigator — Tri-City Medical Center, San Diego, CA; Corey Teigen, MD, Principal Investigator — Sanford Medical Center Fargo, ND
Locations (5):
- United States (5):
  - Tri-City Medical Center, San Diego, California
  - Baptist Health South Florida, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Carolinas Medical Center, Charlotte, North Carolina
  - Sanford Medical Center, Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Mechanical Thrombectomy by the Indigo System: Mechanical Thrombectomy by the Indigo System
Period: Overall Study
Arm/Group | Mechanical Thrombectomy by the Indigo System
Started | 85
Completed | 85
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mechanical Thrombectomy by the Indigo System
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Angiographic Assessment of Vessel Patency at Immediate Post-procedure as Measured by TIMI Scores
Description: Proportion of patients with a post-procedure TIMI score of 2 to 3.
Time Frame: Immediate post-procedure
Population: TIMI score at immediate post-procedure was unavailable for one patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanical Thrombectomy by the Indigo System
Number analyzed (Participants) | 84
Participants | 74

2. Primary Outcome: Procedural Serious Adverse Events
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanical Thrombectomy by the Indigo System
Number analyzed (Participants) | 85
Participants | 5

ADVERSE EVENTS:
Time Frame: up to 24 hours after procedure.
Arm/Group | Mechanical Thrombectomy by the Indigo System
All-Cause Mortality (participants affected / at risk) | 0/85
Serious Adverse Events (participants affected / at risk) | 15/85
Other Adverse Events (participants affected / at risk) | 27/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mechanical Thrombectomy by the Indigo System (N=85)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 1
Intestinal Ischaemia (Gastrointestinal disorders) | 1
Leg Amputation (Surgical and medical procedures) | 2
Myocardial Infarction (Musculoskeletal and connective tissue disorders) | 1
Pulseless Electrical Activity (Cardiac disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Shock (Vascular disorders) | 1
Systemic Inflammatory Response Syndrome (Immune system disorders) | 1
Vascular Pseudoaneurysm Ruptured (Injury, poisoning and procedural complications) | 1
Vessel Puncture Site Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mechanical Thrombectomy by the Indigo System (N=85)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 7
Clostridium Difficule Colitis (Infections and infestations) | 1
Embolism (Vascular disorders) | 5
Epistaxis (Vascular disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Haematuria (Reproductive system and breast disorders) | 1
Haemorrhage (Vascular disorders) | 1
Heparin-Induced Thrombocytopenia (General disorders) | 1
Hypotension (Vascular disorders) | 1
Intestinal Ischaemia (Gastrointestinal disorders) | 1
Leg Amputation (Surgical and medical procedures) | 2
Mental Status Changes (Psychiatric disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pulseless Electrical Activity (Cardiac disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 2
Shock (Cardiac disorders) | 1
Systemic Inflammatory Response Syndrome (Immune system disorders) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Vascular Pseudoaneurysm Ruptured (Injury, poisoning and procedural complications) | 1
Vasospasm (Vascular disorders) | 6
Vessel Puncture Site Haematoma (Vascular disorders) | 1
Visual Impairment (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No